CLINICAL TRIAL: NCT00313742
Title: An Assessment of the Impact of Performing Physical Exercise on the Maximum Plasma Glucose Decline in Subjects With Type 1 Diabetes Managed on a Basal Bolus Insulin Regimen: A Comparison of 3 Basal Insulin Treatments - Insulin Detemir, Insulin Glargine and NPH Insulin
Brief Title: The Effect of Exercise on Blood Glucose Levels in Patients With Type 1 Diabetes: A Comparison of 3 Long-acting Insulins
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN304-1724
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Detemir; Insulin Glargine; Insulin, Isophane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: insulin detemir
Drug: insulin glargine
Drug: insulin NPH

SUMMARY:
This trial is conducted in Europe. The aim of this research is to assess the impact of three basal (long-acting) insulin treatments on blood glucose levels in people with type 1 diabetes when performing physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes
* Current basal-bolus insulin therapy
* HbA1c < 10%
* BMI < 32 kg/m2

Exclusion Criteria:

* Proliferative Retinopathy / Maculopathy
* Recurrent major hypoglycaemias
* Impaired hepatic or renal function
* Cardiac Problems
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-04; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The difference between plasma glucose concentrations immediately pre-exercise and the minimum plasma glucose concentrations (nadir) in the period 0-150 min following exercise | following 4 weeks of treatment

SECONDARY OUTCOMES:
Plasma glucose pre-exercise & post-exercise
Hypoglycaemia episodes (major and minor episodes) during exercise, afterwards & from end of study until 07:30 the following morning
Plasma glucose profile post-exercise
Incidence of adverse events during the trial

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Neuss, Germany
- Newcastle upon Tyne, United Kingdom

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com